CLINICAL TRIAL: NCT05667870
Title: A Lifespan Perspective on Accelerated Aging in Congenital Heart Disease
Brief Title: Accelerated Aging in Newborns and Adults With Congenital Heart Disease
Acronym: AccelerAGE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Collaborators: University Hospital, Ghent (Other); Hasselt University (Other)
Responsible Party: Principal Investigator, Philip Moons, Prof. dr., KU Leuven
Other Study IDs: S66590
Record Dates: First submitted 2022-12-14; First posted 2022-12-29 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Heart Defects, Congenital
Keywords: Congenital heart disease; Aging
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — A peripheral blood sample will be collected from mothers, adult healthy controls (blood donors of the Red Cross) and adults with CHD. For the newborns, only an umbilical cord blood sample will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Newborns with CHD and their mothers: Consecutive newborns with CHD (n=100), who are diagnosed and born in the University Hospitals of Leuven and Ghent, are eligible for inclusion. Mothers (n=100) will be asked for participation in the study before delivery and written informed consent will be obtained. Umbilical cord blood of the ENVIRONAGE study (Hasselt University) will be used as a control group.
- (Young) adults with CHD - study 2: An age-stratified random sample of (young) adults with CHD, followed-up at the University Hospital of Leuven and the Ghent University Hospital will be included. Age strata for this study are: 18-24y; 25-34y; 35-44y; 45-54y; 55+. In total 500 patients will be included, 100 in each age stratum.
- (Young) adults with CHD - study 3: At the University Hospital of Leuven and Ghent University Hospital, patients with selected complex (Fontan operation; Systemic right ventricle), moderate (Tetralogy of Fallot; Coarctation of the aorta), and mild heart defects (isolated atrial septal defect; isolated ventricular septal defect) are eligible. For each type of heart defect 20 patients between the age of 30-50 years are enrolled. The overall sample will comprise 120 patients, who will be part of study 2 as well.
- Healthy controls: Data on healthy controls (n=500) will be retrieved from blood donors at the blood donation service of the Belgian Red Cross-Flanders. The healthy controls will be matched to the included adult patients (in study 2 and 3) based on sex and age.

SUMMARY:
Many childhood-onset diseases used to be lethal. Improved life expectancy yield that most patients can survive into adulthood, to date. However, survivors of childhood-onset diseases often develop morbidities that suggest accelerated aging. Indeed, age-related conditions are observed sooner and more frequently in people with childhood-onset diseases. Congenital heart disease (CHD) is a typical example of a childhood-onset disease and is the most common birth defect, comprising a spectrum of mild, moderate and complex heart defects. Recent studies showed that age-related morbidities occur more often and at an earlier age in these patients. The overall goal of this project is to quantify and understand disparities in chronological and biological age over the lifespan in CHD patients.

DETAILED DESCRIPTION:
Three main research objectives are proposed:

Objective 1: The investigators will determine the biological age in patients with CHD across the lifespan, using established and novel biomarkers for aging, and assess the disparity with chronological age.

Objective 2: The investigators will identify clinical, behavioral, psychological and social predictors of aging in patients with CHD.

Objective 3: The investigators will investigate the difference in biological-chronological age disparity between patients with CHD and healthy counterparts.

Three studies will be performed to investigate these objectives:

Study 1: Newborns with CHD

- The aim is to (i) compare telomere length in newborns with or without CHD; and (ii) to assess pregnancy-related/clinical and mother-related (behavioral, psychological, social) predictors of telomere length in newborns with CHD.

Study 2: (Young) adults with CHD

- This study aims to (i) compare telomere length in age strata of (young) adults with or without CHD; (ii) to assess clinical, behavioral, psychological, and social predictors of telomere length in patients with CHD; and (iii) to explore the relationship with functional outcomes, such as frailty and cognition.

Study 3: Epigenetic clock in adults with CHD

- This study focusses on (i) assessing the biological age by measuring DNA methylation in mild, moderate and complex heart defects, and (ii) determining if the disparity between biological and chronological age is a function of anatomical complexity and functional status of the patients and (iii) comparing the epigenetic clock of adults with and without CHD.

ELIGIBILITY:
1. Newborn with CHD and mother

   Inclusion:
   * Newborns with CHD who are diagnosed and born in UZ Leuven or UZ Gent
   * The mother is able to adequate fill out the questionnaires
   * Informed consent is signed

   Exclusion:
   * The mother does not speak Dutch
   * The heart defect falls within a syndrome condition (e.g., Down syndrome, 22q11 deletion)
   * Very mild heart defects such as a patent foramen ovale, an open ductus of Botalli (no intervention needed), spontaneous closure of ASD/VSD, an isolated mild peripheral pulmonary stenosis
2. Adults with CHD - study 2

   Inclusion:
   * ≥ 18 years of age at the moment of study inclusion
   * Diagnosed with CHD
   * Follow-up at the UZ Leuven or UZ Gent
   * Signed informed consent
   * Physical, cognitive, and language abilities to complete self-report questionnaires/ assessment tests

   Exclusion:
   * Not speaking Dutch
   * Very mild heart defects such as a patent foramen ovale, an open ductus of Botalli (no intervention needed), spontaneous closure of ASD/VSD, an isolated mild peripheral pulmonary stenosis
   * The heart defect falls within a syndrome condition (e.g., Down syndrome, 22q11 deletion)
3. Adults with CHD - study 3

   Inclusion:
   * Included in study 2
   * Between 30-50 years of age at the moment of study inclusion
   * Follow-up at the UZ Leuven or UZ Gent
   * Signed informed consent
   * Physical, cognitive, and language abilities to complete self-report questionnaires/ assessment tests
   * Having one of the following CHD conditions: isolated arterial septal defect, isolated ventricular septal defect, tetralogy of Fallot, coarctation of the aorta, Fontan operation or systemic right ventricle.

   Exclusion
   * Not speaking Dutch
   * The heart defect falls within a syndrome condition (e.g., Downsyndrome, 22q11 deletion)
4. Health volunteers

Inclusion:

* Male or female healthy volunteers of the Red Cross
* Aged 18 - 65 years at the moment of inclusion
* The healthy volunteers must match with the patients included in study 2 based on age and sex
* Signed informed consent
* The requirements of the Red Cross for blood donation are fulfilled

Exclusion:

* Medical history of cardiac, pulmonal, renal or liver disease, chronic anemia, blood clotting disorder
* Not speaking Dutch
* Pregnancy
* Born with a heart condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Newborns with CHD and mother
  2. Adults with CHD - study 2 For each age stratum 100 patients must be included (Gent and Leuven combined), so a total of 500 patients will be included: 18-24 years of age, 25-34 years of age, 35-44 years of age, 45-54 years of age, ≥ 55 years of age
  3. Adults with CHD - study 3 These patients must also be included in study 2. The patients must have the following CHD conditions: isolated arterial septal defect, isolated ventricular septal defect, tetralogy of Fallot, coarctation of the aorta, Fontan operation or systemic right ventricle. Furthermore, they need to be between 30-50 years old.
  4. Healthy volunteers Health volunteers of the Red Cross.
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Telomere length | Baseline
  Telomere length will be measured on umbilical cord blood from newborns and on peripheral blood from adults with and without CHD.

SECONDARY OUTCOMES:
Clinical, behavioral, psychological and social predictors of telomere length | Baseline
  This will be studied by using the life history calendar in adults. In newborns, a pregnancy history calendar and correlation with the maternal telomere length will be used.
Fall history as a functional outcome of aging in adults with CHD | Baseline
  A fall history questionnaire will be used.
Frailty as a functional outcome of aging in adults with CHD | Baseline
  The Fried method is used for assessment of frailty and consists of five parts: self-report questions about unintentional weight loss, exhaustion and physical activity, an assessment of weakness performed using a handgrip dynamometer, and a walk test. A patient is considered non-frail, pre-frail and frail if, respectively, 0, 1-2 or 3/more components are present.
Cognitive impairment as a functional outcome of aging in adults with CHD | Baseline
  The Montréal Cognitive Assessment Screener (MoCA) is used for assessment of cognitive function. The maximum score is 30 points, a score of 26 or higher is considered normal. A lower score indicates a worse cognitive function.
Epigenetic clock in adults with and without CHD | Baseline
  This will be examined based on DNA methylation.
hsCRP in adults with CHD | Baseline
Retina scan in adults with CHD | Baseline
  This will only be performed on patients included in Leuven

CONTACTS AND LOCATIONS:
Overall Officials: Philip Moons, Prof. PhD, Principal Investigator — Professor in Healthcare Sciences
Locations (2):
- Belgium (2):
  - Ghent University Hospital, Ghent
  - University Hospital Leuven, Leuven

IPD SHARING:
Plan to Share IPD: Undecided